CLINICAL TRIAL: NCT05906472
Title: Prevent Unnecessary Surgeon Holds of Ingestions for Tracheostomy (PUSH-IT)
Brief Title: PUSH-IT Continuing Enteral Feeds for Tracheostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Eden Nohra, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY 00005099
Record Dates: First submitted 2023-06-04; First posted 2023-06-18 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Tracheostomy Complication; Critical Illness; Nutritional Deficiency
Keywords: tube feed; nil per os; aspiration; pneumonia; nutritional delivery
MeSH Terms: conditions — Critical Illness; Malnutrition; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Feeds continued (Experimental): Enteral feeds are continued up until time of tracheostomy.
  Interventions: Other: Feeds continued
- Feeds withheld (Other): Enteral feeds are withheld at least 6 hours prior to time of tracheostomy.
  Interventions: Other: Feeds held

INTERVENTIONS:
Other: Feeds continued — Enteral feeds are continued up until time of surgery
  Arms: Feeds continued
Other: Feeds held — Enteral feeds are stopped 6 or more hours before surgery
  Arms: Feeds withheld

SUMMARY:
The goal of this clinical trial is to evaluate nutrition administration in the time around the tracheostomy in patients with breathing tubes. The main questions it aims to answer are:

* Will continuing nutrition up to the time of surgery (tracheostomy) decrease nutrition interruptions, thereby increasing food intake?
* Does continuing nutrition up to the time of surgery increase instances of food going into the lungs or lung infections?

Researchers will compare patients who have nutrition withheld 6 hours prior to surgery versus those who receive nutrition up until the time of surgery to see if there are differences in food intake, instances of food entering the lungs or lung infections.

DETAILED DESCRIPTION:
Malnutrition is a significant problem in the critically ill, however with busy operating room schedules, we often find that feeds are interrupted repetitively prior to elective surgery. These interruptions are practiced based on the American Society of Anesthesiologist guidelines for fasting intervals for elective surgery. These guidelines, however, were not created for critically ill, intubated patients. The theoretical concern for an increased risk of aspiration with continuation of enteral feeds up to the time of surgery persists without supporting evidence. Thus, there is a need for a universal evidence-based guideline on perioperative enteral feeding to benefit critical care patients.

To this end, the goal of the present study is to implement a protocol designed to decrease the interruption of enteral feeds in critical care patients undergoing tracheostomy and prospectively evaluate whether this leads to a quantitative increase in nutritional intake without increasing the risk of aspiration. Additionally, we hope that increasing quantitative nutrition may decrease morbidity especially in the small subset of patients where feed interruptions occur repetitively.

If the aims of the project are achieved, the data obtained from this study will be used to create an evidence-based platform from which physicians can practice. This will end the anecdotal controversy regarding perioperative tube feed management for tracheostomy; thereby increasing quantitative nutrition and hopefully improving the care of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* admitted to the intensive care unit (ICU)
* intubated and require tracheostomy

Exclusion Criteria:

* under 18 years
* unable to obtain informed consent
* deemed clinically brain dead within 7 days of enrollment
* transitioned to comfort measures within 7 days of enrollment
* Pregnant patients
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of aspiration pneumonia | Over 7 days from the time of tracheostomy
  To assess differences in rates of aspiration events, a log-rank test for differences in survival curves model will be used. Assuming proportional hazards and non-informative censoring, a cox-model will be used to estimate follow-up hazard ratios for development of aspiration pneumonia between the two groups of interest.

SECONDARY OUTCOMES:
Volume of tube feed delivery | From day of consent to completion of study which is 7 days from the time of tracheostomy.
  We will compare the volume of tube feeds delivered daily between the two groups for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Marcy Jordan, PhD, Study Director — University at Buffalo
Locations (6):
- United States (6):
  - Nuvance Health - Danbury Hospital, Danbury, Connecticut
  - St. Mary's Medical Center, West Palm Beach, Florida
  - HCA Research Medical Center, Kansas City, Missouri
  - Erie County Medical Center (University at Buffalo), Buffalo, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of South Carolina Sch of Medicine /Prisma Health Richland, Columbia, South Carolina